CLINICAL TRIAL: NCT03310931
Title: Predictive Significance of Thrombelastography on Early Neurological Deterioration in Patients With Acute Ischemic Stroke
Brief Title: Predictive Significance of TEG on END in Patients With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Dongguan People's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhu Shi, MD, Deputy Director of Neurology Department, Dongguan People's Hospital
Other Study IDs: DongguanPeopleH
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — thrombelastography on admission
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- End and non-END groups: END was denied as NIHSS score increase of 2 or more than 2 within 7 days after admission

SUMMARY:
The purpose of this study is to evaluate whether Thromboelastography (TEG) parameters on admission might be predictive for early neurological deterioration in acute ischemic stroke patients, specifically for the DWI lesion evolution within the first week after stroke onset.

DETAILED DESCRIPTION:
Early neurological deterioration (END ) is a major concern in stroke care, consistently associated with adverse clinical outcomes.END is a heterogeneous complex of pathophysiological and clinical entities. Despite some straight forward causes, DWI lesion growth is reportedly a primary underlying mechanism. Early recognition of END risk would allow for timely identification and proper intervention, improving stroke health care.

Thromboelastography (TEG) measures the coagulation process from initial clotting cascade to clot strength, providing an integrated picture of two separate but simultaneously occuring components of coagulation, thrombosis and lysis. It has been reported to be associated with short and long-term outcome in patients with trauma, coronary artery diseases , pulmonary embolism and, most recently, stroke prevention.The purposes of this study is to evaluate how effective TEG is on predicting END, by producing a range of TEG values correlated with clinical and radiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke within 24 hours after symptom onset
* first ever stroke
* give informed consent

Exclusion Criteria:

* receiving thrombolysis
* cardiogenic embolism
* contradiction to serial MRI studies
* taking hemostatic agents (warfarin, oral anticoagulants and etc. )

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes consecutively admitted patients with acute ischemic stroke in Dongguan people's Hospital. Patients would take TEG study within 6 hours after admission, as well as other routine lab tests. Serial MRI studies would be taken on admission and followed up on 7th day afterward, except when patients experience END, in which case followup MRI should be preformed immediately.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
END | fist week after admission
  increase of NIHSS >=2

SECONDARY OUTCOMES:
DWI lesion growth | 7 days
  Large volume or new lesions on followup DWI than the baseline DWI

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan peoples' hospital, Dongguan, Guangdong, China